CLINICAL TRIAL: NCT04670692
Title: Feasibility of Remote Magnetically Controlled Capsule Endoscopy for Upper Gastrointestinal Tract Examination Under Five-generation Network: a Prospective, Open-label, Pilot Trial
Brief Title: Feasibility of Remote MCE for Upper GI Tract Examination Under Five-generation Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5G-MCE
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Gastrointestinal Disease
Keywords: capsule endoscopy, magnetically; 5G network; telemedicine
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5G-MCE examination (Experimental): There will be 20 volunteers assigned to the 5G-MCE system group. These patients will accept the magnetically controlled capsule examination in Yinchuan. After an overnight fasting and drinking 800-1000 mL water and simethicone for gastric dilatation and preparation, the subjects put on the data recorder with the help of the assistant in Yinchuan. Then, the assistant activated the capsule with the capsule locator. The patient is instructed to swallow the capsule with a small amount of water to effectively observe the esophagus and dentate line. After the capsule entering into the stomach, the examination will be performed through the 5G-MCE system by the endoscopist (W.Z.), with experience of more than 1000 cases of MCE operation, in Shanghai.
  Interventions: Other: 5G-MCE examination
- MCE examination (Active Comparator): There will be 20 volunteers assigned to the MCE system group as comparator group. After an overnight fasting and drinking 800-1000 mL water and simethicone for gastric dilatation and preparation, the subjects put on the data recorder with the help of the endoscopist. Then, the endoscopist activated the capsule with the capsule locator. The patient is instructed to assume the left lateral decubitus position and to swallow the capsule with a small amount of water to effectively observe the esophagus and dentate line. Then, under the guidance of the endoscopist (W.Z.) face to face, subject continue the examination of stomach and duodenum.
  Interventions: Other: MCE examination

INTERVENTIONS:
Other: 5G-MCE examination — The endoscopist (W.Z.) manipulated the two joysticks on the remote console (based in Shanghai). Then the remote control software and remote connection software takes the endoscopist's input and translates it into a control signal. After network transmission, the patient side cart (based in Yinchuan) translates the control signal into actual instrument manipulation and mobilize the robotic magnetic arm, and simultaneously driving the precise movement and rotation of the capsule to perform the gastric and duodenum examination. Meanwhile, the images captured by the capsule are simultaneously sent back to the screen of the remote console, and thus provide guidance for better control of the capsule.
  Arms: 5G-MCE examination
Other: MCE examination — The endoscopist (W.Z.) performs the MCE examination procedure conventionally. And communicate with the volunteer face to face in the same examination room.
  Arms: MCE examination

SUMMARY:
With the combination of robotic and 5G network communication technology, telemedicine becomes more and more feasible and efficient. Magnetically controlled capsule endoscopy (MCE) has been confirmed to have comparable accuracy with conventional gastroscopy with the advantages of comfort and convenience. 5G communication technology has been applied to several fields in telemedicine, but its effectiveness, safety, and stability in remote magnetically controlled capsule endoscopy for upper gastrointestinal tract examination have not been established. The aim of this study is to evaluate the diagnostic utility, safety, feasibility and patient's acceptability of remote magnetically controlled capsule endoscopy system under 5G network.

DETAILED DESCRIPTION:
With the combination of robotic and 5G network communication technology, telemedicine becomes more and more feasible and efficient. On the one hand, telemedicine can conserve and optimize medical resources, providing high-quality medical services to unbalanced areas, such as rural areas, stricken areas and battlefields. On the other hand, telemedicine can reduce the time spent by patients waiting for examination and treatment and thus prevent diseases from worsening.

Magnetically controlled capsule endoscopy (MCE) has been confirmed to have comparable accuracy with conventional gastroscopy with the advantages of comfort and convenience. 5G communication technology has been applied to several fields in telemedicine, but its effectiveness, safety, and stability in remote magnetically controlled capsule endoscopy for upper gastrointestinal tract examination have not been established.

The 5G-MCE system was provided by Ankon Technologies Co, Ltd (Shanghai, China), this system consists of three parts: remote console, remote control software (NaviRemoteCtrl), and remote connection software (NaviRemoteConn). The remote console (based in Shanghai), takes the endoscopist's input and translates it into a control signal. After network transmission, the patient side cart (based in Yinchuan) translates the control signal into actual instrument manipulation. The images captured by the capsule are simultaneously sent back to the screen of the remote console, and thus provide guidance for better control of the capsule.

The aim of this study is to evaluate the diagnostic utility, safety, feasibility and patient's acceptability of remote magnetically controlled capsule endoscopy system under 5G network.

ELIGIBILITY:
Inclusion Criteria:

1. Gender is not limited.
2. Patients aged 18 years or older.
3. Both inpatients and outpatients.
4. Volunteers with or without abdominal complaints.
5. Able to provide informed consent.

Exclusion Criteria:

1. dysphagia or symptoms of gastric outlet obstruction, suspected or known intestinal stenosis,overt gastrointestinal bleeding,fistulas and strictures;
2. history of upper gastrointestinal surgery or suspected delayed gastric emptying;
3. Patients with poor general condition,asthma or claus trophobia;
4. Implanted metallic devices such as pacemakers,defibrillators, artificial heart valves or joint prostheses;
5. Pregnancy or mentally ill person;
6. currently participating in another clinical study;
7. communication obstacles persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Maneuverability score | During the procedure
  Maneuverability score was the sum of four subjective scores rated by the operator (signal transmission quality score, operating comfort score, gastric visualization score and study subject compliance score), each of which ranged from 1 to 5 denoting the lowest to the highest degree of satisfaction.

SECONDARY OUTCOMES:
Gastric examination time(GET) | During the procedure
  GET was defined as the time time taken for the endoscopist to complete the gastric examination to his or her satisfaction.
the comfort and acceptability of patients | After the procedure(within 5 days)
  The investigators use a satisfaction questionnaire to evaluate the comfort and acceptability of each patient
diagnostic yield | after the procedure(within 5 days)
  Diagnosis based on the data of 5G-MCE by two endoscopist
Adverse events | During and within 2 weeks after the procedure
  Adverse events during and after the procedure
Clinical success | During the procedure
  Complete observation of the mucosa (>90% of the mucosa observed) in gastric cardia, fundus, body, angulus, antrum and pylorus.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liao Z, Duan XD, Xin L, Bo LM, Wang XH, Xiao GH, Hu LH, Zhuang SL, Li ZS. Feasibility and safety of magnetic-controlled capsule endoscopy system in examination of human stomach: a pilot study in healthy volunteers. J Interv Gastroenterol. 2012 Oct-Dec;2(4):155-160. doi: 10.4161/jig.23751. Epub 2012 Oct 1. PMID 23687601
- [Background] Zou WB, Hou XH, Xin L, Liu J, Bo LM, Yu GY, Liao Z, Li ZS. Magnetic-controlled capsule endoscopy vs. gastroscopy for gastric diseases: a two-center self-controlled comparative trial. Endoscopy. 2015 Jun;47(6):525-8. doi: 10.1055/s-0034-1391123. Epub 2015 Jan 15. PMID 25590177
- [Background] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- [Background] Qian YY, Zhu SG, Hou X, Zhou W, An W, Su XJ, McAlindon ME, Li ZS, Liao Z. Preliminary study of magnetically controlled capsule gastroscopy for diagnosing superficial gastric neoplasia. Dig Liver Dis. 2018 Oct;50(10):1041-1046. doi: 10.1016/j.dld.2018.04.013. Epub 2018 Apr 24. PMID 29779696
- [Background] Zhao AJ, Qian YY, Sun H, Hou X, Pan J, Liu X, Zhou W, Chen YZ, Jiang X, Li ZS, Liao Z. Screening for gastric cancer with magnetically controlled capsule gastroscopy in asymptomatic individuals. Gastrointest Endosc. 2018 Sep;88(3):466-474.e1. doi: 10.1016/j.gie.2018.05.003. Epub 2018 May 9. PMID 29753039
- [Background] Chen X, Gao F, Zhang J. Screening for Gastric and Small Intestinal Mucosal Injury with Magnetically Controlled Capsule Endoscopy in Asymptomatic Patients Taking Enteric-Coated Aspirin. Gastroenterol Res Pract. 2018 Nov 15;2018:2524698. doi: 10.1155/2018/2524698. eCollection 2018. PMID 30581462
- [Background] Zhu SG, Qian YY, Tang XY, Zhu QQ, Zhou W, Du H, An W, Su XJ, Zhao AJ, Ching HL, McAlindon ME, Li ZS, Liao Z. Gastric preparation for magnetically controlled capsule endoscopy: A prospective, randomized single-blinded controlled trial. Dig Liver Dis. 2018 Jan;50(1):42-47. doi: 10.1016/j.dld.2017.09.129. Epub 2017 Oct 6. PMID 29110963
- [Background] Wang YC, Pan J, Jiang X, Su XJ, Zhou W, Zou WB, Qian YY, Chen YZ, Liu X, Yu J, Yan XN, Zhao AJ, Li ZS, Liao Z. Repetitive Position Change Improves Gastric Cleanliness for Magnetically Controlled Capsule Gastroscopy. Dig Dis Sci. 2019 May;64(5):1297-1304. doi: 10.1007/s10620-018-5415-7. Epub 2018 Dec 17. PMID 30560329
- [Background] Jiang X, Qian YY, Liu X, Pan J, Zou WB, Zhou W, Luo YY, Chen YZ, Li ZS, Liao Z. Impact of magnetic steering on gastric transit time of a capsule endoscopy (with video). Gastrointest Endosc. 2018 Oct;88(4):746-754. doi: 10.1016/j.gie.2018.06.031. Epub 2018 Jul 11. PMID 30005825
- [Background] Li JO, Liu H, Ting DSJ, Jeon S, Chan RVP, Kim JE, Sim DA, Thomas PBM, Lin H, Chen Y, Sakomoto T, Loewenstein A, Lam DSC, Pasquale LR, Wong TY, Lam LA, Ting DSW. Digital technology, tele-medicine and artificial intelligence in ophthalmology: A global perspective. Prog Retin Eye Res. 2021 May;82:100900. doi: 10.1016/j.preteyeres.2020.100900. Epub 2020 Sep 6. PMID 32898686
- [Background] Hong Z, Li N, Li D, Li J, Li B, Xiong W, Lu L, Li W, Zhou D. Telemedicine During the COVID-19 Pandemic: Experiences From Western China. J Med Internet Res. 2020 May 8;22(5):e19577. doi: 10.2196/19577. PMID 32349962
- [Background] Zheng J, Wang Y, Zhang J, Guo W, Yang X, Luo L, Jiao W, Hu X, Yu Z, Wang C, Zhu L, Yang Z, Zhang M, Xie F, Jia Y, Li B, Li Z, Dong Q, Niu H. 5G ultra-remote robot-assisted laparoscopic surgery in China. Surg Endosc. 2020 Nov;34(11):5172-5180. doi: 10.1007/s00464-020-07823-x. Epub 2020 Jul 22. PMID 32700149
- [Derived] Zhang T, Chen YZ, Jiang X, He C, Pan J, Zhou W, Hu JP, Liao Z, Li ZS. 5G-based remote magnetically controlled capsule endoscopy for examination of the stomach and small bowel. United European Gastroenterol J. 2023 Feb;11(1):42-50. doi: 10.1002/ueg2.12339. Epub 2022 Nov 23. PMID 36416805